CLINICAL TRIAL: NCT04489212
Title: A Study of Mucosal Sparing Adjuvant Radiotherapy After Surgical Exploration in HPV + Head and Neck Cancer of Unknown Primaries (HNCUP)
Brief Title: Study of Mucosal Sparing Adjuvant Radiotherapy After Surgical Exploration in HPV+ Head and Neck Cancer of Unknown Primaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1974; NCI-2020-05152 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1974 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Head and Neck Carcinoma of Unknown Primary; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (follow-up, observation) (Experimental): Patients who have recurrence or progression during treatment or observation have medical charts are reviewed every 6 months for 5 years. Patients who complete adjuvant treatment are followed for observation 3 days after radiation therapy, 1 month after radiation therapy, every 3 months after radiation therapy for 2 years, every 6 months for 1 year, and then annually for 2 years.
  Interventions: Other: Medical Chart Review; Other: Patient Observation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the clinical outcome of mucosal sparing adjuvant radiotherapy after surgical exploration in HPV+ head and neck cancer of unknown primaries. The purpose of this research is to assess if radiation treatment to the neck only for tumors with unclear original locations after careful surgical evaluation will lead to historical rates of disease control while reducing side effects and toxicity from treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the rate of manifestation of an occult primary tumor in the pharyngeal axis or delayed nodal recurrence in a un-dissected and/or non-irradiated neck at 2 years after study registration in patients treated with mucosal sparing (and unilateral neck, if applicable) radiotherapy after resection using transoral surgery for head and neck cancer of unknown primaries (HNCUP).

SECONDARY OBJECTIVES:

I. To describe the rates and severity of acute and late toxicities and PEG dependence attributable to mucosal sparing radiotherapy after resection using transoral surgery by assessment of grade 3 or higher adverse events National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0 criteria.

II. To describe the overall survival, recurrence-free survival (manifestation of an occult primary in the pharyngeal axis, nodal recurrence in a treated (surgery/radiation therapy [RT]) neck, delayed lymph node metastasis in an untreated neck (surgery/RT), and distant failure associated with mucosal sparing radiotherapy.

III. To describe swallowing function changes (assessed via swallowing study) associated with transoral surgery and adjuvant mucosal sparing radiotherapy.

OUTLINE:

Patients who have recurrence or progression during treatment or observation have medical charts reviewed every 6 months for 5 years. Patients who complete adjuvant treatment are followed for observation 3 days after radiation therapy, 1 month after radiation therapy, every 3 months after radiation therapy for 2 years, every 6 months for 1 year, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients meet criteria for intensity-modulated proton therapy (IMPT) treatment for oropharyngeal cancer

  * If IMPT is declined by patient's insurance, they can be treated with standard of care IMRT using the same applicable standard of care procedures outlined in the procedures manual
* Meet criteria for adjuvant chemotherapy (if applicable)
* Histological confirmation of human papillomavirus (HPV)+ squamous cell carcinoma as defined by neck node pathology. HPV positivity will be defined as positive staining for p16 and HPV deoxyribonucleic acid (DNA) in situ hybridization (ISH). (If discordant, ribonucleic acid [RNA] ISH will be run for confirmatory testing)
* Clinical stage T0 N1-N3 and confirmed pathologic stage T0 N1-N2 M0 (American Joint Committee on Cancer [AJCC] 8th edition) with one of the following risk factors:

  * Lymph node >= 3 cm
  * >= 2 positive lymph nodes
  * Presence of extracapsular extension
  * > 1 nodal level involved
* Absence of distant metastases on standard diagnostic workup, prior to registration (chest computed tomography [CT], chest x-ray [CXR], or positron emission tomography [PET]/CT)
* Able to undergo pre-operative Q-clear series PET/CT head/neck for diagnostic workup of occult primary and nodal disease
* Able to undergo transoral surgery and neck dissection by their ears, nose, and throat (ENT) oncologist

  * Surgical exploration/sampling of all mucosal sites including ipsilateral wide field tonsillectomy and base of tongue resection. Additional biopsies or surgical excision at the surgeon's discretion. Any radiographic or clinically suspicious areas should be biopsied or removed. Bilateral neck dissection for high risk patients. Ipsilateral dissection only, for patients with contralateral cN0 necks and negative preoperative imaging
  * Final pathologic evaluation demonstrating all benign samplings without discernible primary
* Documented smoking history
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 35 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 35 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 35 days prior to registration)
* Creatinine =< 1.5 mg/dL or creatinine clearance >= 50 mL/min (obtained =< 35 days prior to registration)
* Total or direct bilirubin < 2 x institutional upper limit of normal (ULN) (obtained =< 35 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 x institutional ULN (obtained =< 35 days prior to registration)
* Ability to complete questionnaire(s) by themselves or with assistance
* Able to provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any patient with positive retropharyngeal nodes on imaging
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other active malignancy =< 5 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer, breast cancer, prostate cancer, well-differentiated thyroid cancer, carcinoma-in-situ of the cervix. NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of connective tissue disorders such as scleroderma, rheumatoid arthritis, lupus, or Sjogren's disease
* Prior history of radiation therapy to the affected site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Primary local recurrence | At 2 years
  Will be estimated by counting up the number of patients with an occult primary tumor within the pharyngeal axis or nodal recurrence in untreated neck and dividing by the total number of eligible patients.

SECONDARY OUTCOMES:
Incidence of acute grade 3 or higher functional mucosal adverse events | Up to 1 month post radiation therapy (XRT)
  Will characterize the acute grade 3 or higher functional mucosal adverse events (up to 1 month post-XRT) associated with mucosal sparing.
Overall survival (OS) | From registration to death due to any cause, assessed up to 5 years
  The distribution of OS will be estimated using the method of Kaplan-Meier.
Recurrence-free survival (RFS) | From registration to the first of either disease recurrence, delayed lymph node metastasis in an untreated neck (contralateral), development of distant metastatic disease, or death, assessed up to 5 years
  The distribution of RFS will be estimated using the method of Kaplan-Meier.
Distant metastasis rates | Up to 2 years
Change in swallowing function | Up to 5 years
  To describe swallowing function changes (assessed via swallowing study) associated with transoral surgery and adjuvant mucosal sparing radiotherapy. Swallowing will be scored (yes, no) for aspiration, penetration, velopharyngeal incompetence, epiglottic eversion, tongue base retraction, and pharyngeal swallow response using the metric outlined by Eisbruch et al. Swallowing assessments will be completed at baseline, along with 3 and 12 months after the completion of protocol XRT. The swallowing questions will be explored descriptively to detect patterns and substantial changes over time. In addition, McNemar's tests (or Wilcoxon signed-rank tests) for paired samples will be used to see if the swallowing questions significantly change over time for each post-baseline time point. MBSImp scoring and the Penetration/aspiration scale scores will be assessed as well.
Incidence of acute adverse events | Up to 1 month post-XRT
  The maximum grade for each type of acute adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns, especially focusing on grade 3+ adverse events, regardless of attribution to the study treatment.
Incidence of late adverse events | Up to 2 years post-XRT
  The maximum grade for each type of adverse event will be recorded for each patient for up to 2 years post-treatment, and frequency tables will be reviewed to determine patterns, especially focusing on grade 3+ non-hematologic adverse events, regardless of attribution to the study treatment. Hematologic adverse events will not be followed closely long-term given that adjuvant treatment is only given for 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Ma, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials